CLINICAL TRIAL: NCT00382785
Title: Psychosocial Outcomes in Online Cancer Support Groups
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Paula Klemm, PhD, RN, OCN, University of Delaware School of Nursing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DDD#504604
Record Dates: First submitted 2006-09-28; First posted 2006-10-02 (Estimated); Results first posted 2010-12-21 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-11

CONDITIONS: Breast Cancer
Keywords: online; support; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- moderated online support (Experimental): 12-week online support led by a healthcare professional
  Interventions: Behavioral: moderated support
- peer-led support (Experimental): 12-week online support group in a peer-led format
  Interventions: Behavioral: peer-led

INTERVENTIONS:
Behavioral: moderated support — one 12-week online support group led by a professional healthcare provider
  Arms: moderated online support
Behavioral: peer-led — 12-week online support in a peer-led format
  Arms: peer-led support

SUMMARY:
Purpose: The purpose of this project is to evaluate whether psychosocial outcomes in women with breast cancer differ based on the format of online group support. This objective will be addressed by the following specific aims:

1. Specific Aim #1 is to determine if there is a difference in depressive symptoms between women with breast cancer assigned to one of two treatment conditions: moderated online support or peer-led online support.

   • H1: Women with breast cancer who participate in moderated online support will report fewer depressive symptoms than women with breast cancer in peer led online support.
2. Specific Aim #2 is to determine if there is a difference in perceived social support between women with breast cancer who are assigned to one of two treatment conditions: moderated online support or peer-led online support.

   • H2: Women with breast cancer who participate in moderated online support will report greater perceived social support than women with breast cancer in peer-led online support.
3. Specific Aim #3 is to determine if there is a difference in quality of life in women with breast cancer who are assigned to one of two treatment conditions: moderated online support or peer-led online support.

   * H3: Women with breast cancer who participate in moderated online support will report better quality of life than women with breast cancer in peer-led online support.

NOTE: Once the study began, it was obvious that we could not prevent anyone from joining a support group, if that was her choice. We also could not control if participants joined a second online support group or face-to-face group during the study. Therefore, we decided to omit a "usual care" (no support) group. The study was completed with just two groups: moderated and peer-support.

DETAILED DESCRIPTION:
Purpose/Specific Aims: The purpose of this randomized two-group longitudinal study is to evaluate whether psychosocial outcomes in women with breast cancer differ based on the format of online group support. Rationale/Significance of study: No research has explored differences in psychosocial outcomes between online support groups that use a professional moderator and those that use a peer-led (self-help) format. This study will address one of the goals put forth in the 2003-2005 ONS Research Agenda, by studying the effects of technology based interventions (online support) on psychosocial outcomes (depression, perceived social support, quality of life) in women with breast cancer. This work will add to the nursing research base with regard to online support for women with breast cancer and provide a springboard for additional studies to enhance the research base. Conceptual Framework: The concept of openness, based on the mutual interaction between human beings and their environment, and emphasized in Rogers' Science of Unitary Human Beings provides a basis for this project. The research will utilize two different support environments and measure how interactions in each affect psychosocial outcomes over time. Main Research Variables: The independent variables are two treatment conditions (moderated online support, peer-led online support). The dependent variables are depressive symptoms, perceived social support, and quality of life. Design: A randomized longitudinal design, comparing two types of online support groups, on the basis of three principal measures, will be used. Each measure will be obtained at baseline and at three later timepoints. Setting: Support groups will be accessed from secure and password protected university web pages devoted exclusively to this study. Sample: Sixty women with breast cancer, at least 21 years of age, who have Internet access will be recruited. Methods: Women will be randomly assigned to one of the two treatment conditions (moderated online support, peer-led online support) given a password, and instructed to complete a Demographic Form and the study questionnaires online. All subjects will be asked to complete the study questionnaires again at 6, 12, and 16 weeks. Moderated groups will run in a semi-structured format over 12 weeks, with a different discussion topic moderated each week by the moderator. Peer-led groups will be run in a peer support format over 12 weeks. Implications for practice: Women with breast cancer are turning to online resources for support. Nurses should be aware of the benefits/limitations of this support alternative. A cost benefit may be suggested if it is shown that peer-led online support has psychosocial benefits similar to professionally facilitated groups. Additional research is needed to explore the impact of online support on psychosocial outcomes in people with other cancers, minorities, and men. This study will add important information to the research base regarding online support groups and help determine the best strategy for online cancer support.

NOTE: It was obvious that we could not prevent anyone from joining a support group, if that was her choice. We also could not control if participants joined a second online support group or face-to-face group during the study. Therefore, we dropped the "usual care" (no support) group. The study was completed with just two groups: moderated and peer-support.

ELIGIBILITY:
Inclusion Criteria: Clinical diagnosis of breast cancer

* Female
* At least 21 years of age
* Internet access; Able to read and write English
* Have completed treatment for breast cancer in the past 36 months or are receiving treatment
* Do not currently belong to an online or face-to-face cancer support group
* Internet access

Exclusion Criteria:

* Male
* not diagnosed with breast cancer
* under 21 years of age
* received treatment more than 36 months ago for breast cancer
* no Internet access
* unable to read and write English

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paula Klemm, PhD, Principal Investigator — University of Delaware School of Nursing
Locations (1):
- University of Delaware, Newark, Delaware, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited via flyers, word of mouth, at clinics, and via university electronic news. Participants were recruited from August 2005 through December 2008.
Groups:
- Moderated Group: one 12-week online support group led by a professional healthcare provider
- Non-facilitated (Peer-led): 12-week online support in a peer-led format
Period: Overall Study
Arm/Group | Moderated Group | Non-facilitated (Peer-led)
Started | 25 | 26
Completed | 25 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderated Group | Non-facilitated (Peer-led) | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 25 | 48
  >=65 years | 2 | 1 | 3
Age Continuous [Mean (Standard Deviation); unit: years] | 52.97 (10.75) | 51.52 (8.92) | 52.25 (9.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Personal Resource Questionnaire 85.
Description: The Personal Resource Questionnaire 85 (PRQ85), Part II measures perceived social support and consists of 25 items in a seven-point Likert format which are rated from seven (7) strongly agree, to one (1) strongly disagree. Scores range from 25 to 175 with higher scores indicative of higher levels of perceived social support. Alpha reliability of the PRQ 85 has been demonstrated at >.90
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Moderated Group | Non-facilitated (Peer-led)
Number analyzed (Participants) | 25 | 26
Scores on a scale | 50.22 (3.23) | 53.44 (3.08)
Statistical Analysis 1: Comparison: Moderated Group vs Non-facilitated (Peer-led); Power calculation indicated that 60 subjects would be needed. Null Hypothesis: There will be no difference in perceived social support based on type of online support group (moderated or peer-led); Test type: Superiority or Other; p = .315, univariate analysis

2. Primary Outcome: Scores on the CES-D Scale
Description: The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20-item self-report scale widely used in the assessment of depression. Each item is given a rating of 0 to 3, with a potential range of 0 to 60 for the entire scale. Higher scores are associated with depression. The cutoff for the diagnosis of Major Depressive Disorder on the CES-D is 16. The instrument is a reliable measure (Alpha >.85) of depression
Time Frame: 16 weeks
Population: Same as number of participants analyzed
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Moderated Group | Non-facilitated (Peer-led)
Number analyzed (Participants) | 25 | 26
Scores on a scale | 9.65 (1.98) [-5.77 to 12.21] | 12.97 (1.84) [-12.21 to 5.77]
Statistical Analysis 1: Comparison: Moderated Group vs Non-facilitated (Peer-led); Power analysis indicated that 60 subjects were needed. Null hypothesis: There will be no difference in depressive symptoms based on type of online support group (moderated or peer-led); Test type: Superiority or Other; p = .23, univariate analysis; Null Hypothesis: There will be no difference between the moderated and peer-led groups based on type of online support (moderated; peer-led)

3. Primary Outcome: Scores on the Quality of Life (QOL) Question on the Rotterdam Symptom Check List (RSCL).
Description: The Rotterdam Symptom Checklist (RSCL) measures quality of life in cancer patients. The RSCL checklist includes a QOL life question on a scale of 1 (excellent) to 7 (extremely poor). This was used as a measure of overall QOL.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Moderated Group | Non-facilitated (Peer-led)
Number analyzed (Participants) | 25 | 26
Scores on a scale | 1.90 (.31) [-2.92 to 5.43] | 2.30 (.36) [-5.43 to 2.92]
Statistical Analysis 1: Comparison: Moderated Group vs Non-facilitated (Peer-led); Power analysis indicated that 60 subjects were needed. Null hypothesis: There will be no difference in quality of life (QOL) based on type of online support group (moderated or peer-led); Test type: Superiority or Other; p = .32, Univariate Analysis

ADVERSE EVENTS:
Groups:
- Peer-led: peer-led group
Arm/Group | Moderated | Peer-led
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 0/25 | 0/26

LIMITATIONS AND CAVEATS:
One limitation was the lack of a control group of women who did not take part in an online or face-to-face support group. The reasons for this are explained above.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No